CLINICAL TRIAL: NCT05058807
Title: Effects of Whole Body Vibration on Balance, Strength, Glycosylated Hemoglobin Levels in Diabetic Peripheral Neuropathy
Brief Title: Effects of Whole Body Vibration in Diabetic Peripheral Neuropathy .
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Quratulain
Record Dates: First submitted 2021-09-17; First posted 2021-09-28 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Diabetic Neuropathies
MeSH Terms: conditions — Diabetic Neuropathies

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Whole body vibration group (Experimental): Experimental Group will receive WBV training and balance exercises under the supervision of a physical therapist by using a vibration platform. Balance exercises include:
  Double leg stance with eyes open and eyes closed 10 Reps * 3 minutes Tandem walk for 3 minutes Sideways walk for 3 minutes Single leg stance for 1 minute with 5 Reps, with 30 sec rest interval
  WHOLE BODY VIBRATION:
  The patient stood on the platform with his/her feet barefoot shoulder width and stared at the front, delivered on a side alternating vibration platform in an intermittent way: five repetitions of 1 min vibration followed by a 1 min rest. The vibration frequency and amplitude were 20 Hz and 3.0 mm respectively.
  These outcomes will be evaluated at baseline, and after 4 week and at 8th week
  Interventions: Other: Whole body vibration group
- TAI CHI Group (Active Comparator): Control group will receive Balance exercises include:
  Double leg stance with eyes open and eyes closed 10 Reps * 3 minutes Tandem walk for 3 minutes Sideways walk for 3 minutes Single leg stance for 1 minute with 5 Reps ,with 30 sec rest interval Yang style Tai chi exercise which consist of 10 positions.
  1. Hold the ball ward off 2: Grasping the sparrows tail left; 3.Grasping the sparrows tail Right;; 5.Repulse Monkey; 6. Part wild horse's Mane; 7.Brush knee Twist step; 8.Lift kick left;
  .Lift kick Right; 10.Cross hands with double leg stance
  1st and 2nd week will last for 5reps, 3rd and 4th week will last for 10reps,5th and 6th week will last for 15reps,7th and 8th week will last for 20reps, starting with 10 minutes warming- up and ending with 10 minutes cool-down. These outcomes will be evaluated at baseline, and after 4 week and at 8th week.
  Interventions: Other: Tai Chi group

INTERVENTIONS:
Other: Whole body vibration group — Experimental Group will receive WBV training and balance exercises under the supervision of a physical therapist by using a vibration platform. Balance exercises include:
  Double leg stance with eyes open and eyes closed 10 Reps * 3 minutes Tandem walk for 3 minutes Sideways walk for 3 minutes Single leg stance for 1 minute with 5 Reps, with 30 sec rest interval
  WHOLE BODY VIBRATION:
  The patient stood on the platform with his/her feet barefoot shoulder width and stared at the front, delivered on a side alternating vibration platform in an intermittent way: five repetitions of 1 min vibration followed by a 1 min rest. The vibration frequency and amplitude were 20 Hz and 3.0 mm respectively.
  These outcomes will be evaluated at baseline, and after 4 week and at 8th week
  Arms: Whole body vibration group
Other: Tai Chi group — Control group will receive Balance exercises include:
  Double leg stance with eyes open and eyes closed 10 Reps * 3 minutes Tandem walk for 3 minutes Sideways walk for 3 minutes Single leg stance for 1 minute with 5 Reps ,with 30 sec rest interval Yang style Tai chi exercise which consist of 10 positions. 1. Hold the ball ward off 2: Grasping the sparrows tail left; 3.Grasping the sparrows tail Right;; 5.Repulse Monkey; 6. Part wild horse's Mane; 7.Brush knee Twist step; 8.Lift kick left; 9.Lift kick Right; 10.Cross hands with double leg stance
  1st and 2nd week will last for 5reps, 3rd and 4th week will last for 10reps,5th and 6th week will last for 15reps,7th and 8th week will last for 20reps, starting with 10 minutes warming- up and ending with 10 minutes cool-down. These outcomes will be evaluated at baseline, and after 4 week and at 8th week
  Arms: TAI CHI Group

SUMMARY:
The aim of this study is to conduct a randomized controlled trail to compare and analyze the effects of both whole body vibrator (WBV) and Tai Chi program on static and dynamic postural balance variables of the diabetic population. The purpose of the study is to determine that whether whole body vibrator is more evident for promoting functional independency and improving balance in diabetic neuropathy. Hence distinguishing choices to prevent fall and advancing functional independency by using the appropriate intervention without using extreme loads.

DETAILED DESCRIPTION:
Diabetes Mellitus (DM) is defined as a state of hyperglycemia, in either fasting or postprandial states. DM is a group of metabolic diseases characterized by hyperglycemia resulting from defects in insulin secretion, insulin action, or both . Type 2 diabetes mellitus (T2DM) is one of these diseases and it is characterized by insulin resistance . The International Diabetes Federation (IDF) estimates that the global prevalence of diabetes mellitus is 366 million in 2011 and expects an increase to 552 million in 2030. In this sense, the increase in the DM prevalence, especially in T2D, has become one of the major problems in modern society [5]. In this regard, this chronic disease is connected with the increase of obesity prevalence [6] and the high levels of physical inactivity [5] in people with T2DM.

Peripheral neuropathy is one of the most common complications and consequences of chronic hyperglycemia . This is characterized by a progressive degeneration that primarily affects the small-diameter cutaneous nociceptive fibers. Diabetic patients encounter impaired balance, proprioception loss and decreased ROM. Physical exercise has become a therapy for people with T2DM , improving physical fitness , quality of life, and autonomic modulation ; as well as enhancing metabolic control and insulin sensitivity; and reducing inflammatory markers and neuropathy symptoms . Interestingly, physical activity could also increase the regenerative capacity of cutaneous axons, slowing or preventing neuropathy progression .

Exercises based on whole-body vibration (WBV) training have shown to enhance balance, mobility muscle strength, pain, cardiorespiratory fitness, and bone density, in both healthy and clinical populations. In this regard, a recent systematic review and meta-analysis (with a total of seven studies, involving 279 older adults with T2DM) focused on the effects of WBV determined that this training improved the mobility, balance and aerobic capacity without any known adverse effects. Moreover, WBV could have positive effects on glycemic indices or body composition. Regarding glycemic indices, a previous study showed that acute WBV decreases the glucose level in elderly women with T2DM. However, the effects of WBV intervention on glycosylated hemoglobin (HbA1c) is uncertain. Tai Chi exercise program which is actually a form of proprioceptive and balance training helps in reduction of fall and balance issues and also beneficial for the pain reduction in osteoarthritic patients.

Basic TC exercise is a mind-body exercise composed of a series of refined motions linked together as a rhythmical sequence in which the body is continuously shifting with low center of gravity from one foot to the other. These exercises can help in training of dual task performance as the practitioner's eye focuses on the leading arm and the mind focuses on the breath and movement sequences. It also improves cardiovascular endurance, aerobic capacity and quality of life and reduces stress

ELIGIBILITY:
Inclusion Criteria:

* Balance : 21-52
* DM type II from past 10 years
* American Diabetes Association (ADA) guideline 2001 or using oral hypoglycemic agent; HbA1C < 8.5 %
* Taking Medicine and stable patients
* MMSE>25
* Michigan Diabetic Neuropathy Score (MDNS) between 13 and 29 (mild to moderate neuropathy)

Exclusion Criteria:

* Patients with any musculoskeletal impairment (such as inability to walk independently), vision impairment, vestibular diseases with a diabetes-related etiology, or dementia (Mini-Mental State Examination score < 24/30)

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
•Berg Balance Scale | Change from Baseline mobility and balance to 4th week, 8 Weeks
  BBS is a gold standard tool, developed by Berg et al. in 1998 for functional assessment of balance. It has been widely used for older people with balance impairments, stroke, Parkinson's disease, vestibular disorders and in different healthcare settings (7,23). It consists of 14 items to detect static (5 items) and dynamic (9 items) balance. Each item has a score of 0-4 on ordinal scale. Total score is 56, higher the score better is the balance. 0-20 indicates poor balance and predicts high risk of fall, 21-40 indicates acceptable balance and medium fall risk and 41-56 indicates good balance and low fall risk (7, 24). BBS exhibits an excellent reliability; test-retest (ICC) = 0.91) and inter-rater (ICC = 0.97). This scale also has some limitations such as it has a little focus on gait and dynamic balance. Secondly, it has ceiling effect that was reported as 22.5% in community-dwelling older adults
5 times sit to stand test | Change from Baseline balance to 4th week ,8th Weeks
  To evaluate lower-limb muscle strength, the five-times-sit-to stand (FTSTS) test was used. For this test, the subject was asked to sit in an armless chair (with its back supported against a wall) with arms crossed over his/her chest and then instructed to stand and sit five times as quickly as possible. The same chair was used for all subjects. Subjects performed two timed trials. The instructor commenced the test with "Ready, Set, Go", started a digital stopwatch on "Go," and counted aloud each of the five completed sit to stand cycles. The stopwatch was stopped when the subject returned to the seated position for the fifth time

SECONDARY OUTCOMES:
Single leg stance test | Change from Baseline , balance and fall prevention to 4Weeks, 8 weeks
  The Single leg Stance (SLS) Test is used to assess static postural and balance control. Balance assessments (like SLS test) are a valuable clinical tool for monitoring neurological and musculoskeletal status as well as for managing fall risk

CONTACTS AND LOCATIONS:
Overall Officials: Misbah ghous, MS, Principal Investigator — Riphah International University Islamabad
Locations (1):
- Pakistan General Railway Hospital, Rawalpindi, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No